CLINICAL TRIAL: NCT03724955
Title: Pilot Study Evaluating the Effects of Estradiol for Hypogonadal Women With Cystic Fibrosis and Osteopenia
Brief Title: Pilot E2 for Hypogonadal Women With CFBD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Issues with Recruitment.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Vin Tangpricha, MD, PH.D, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00107135
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Cystic Fibrosis Related Bone Disease
Keywords: Hypogonadism; Estrogen Supplement
MeSH Terms: conditions — Hypogonadism | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded, randomized, placebo-controlled, interventional
Who Masked: Participant, Outcomes Assessor
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Group (Experimental): The treatment group will receive Estradiol 2 mg oral daily for 6 months. Medication will be mailed to patient. All study drugs will be dispensed by the Investigational Drug Pharmacy.
  Interventions: Drug: Estradiol 2 mg
- Placebo Group (Placebo Comparator): The placebo group will receive placebo oral daily for 6 months. Medication will be mailed to patient. Placebo will be dispensed by the Investigational Drug Pharmacy.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Estradiol 2 mg — Participants in this arm will receive Estradiol 2 mg oral daily for 6 months
  Other Names: Estrace
  Arms: Treatment Group
Other: Placebo — The placebo group will receive placebo oral daily for 6 months
  Arms: Placebo Group

SUMMARY:
The study is a prospective, double blinded, placebo controlled, randomized study to evaluate the effects of daily oral estrogen supplements on bone health, sexual and reproductive health, quality of life and markers of inflammation and lung function when given to hypogonadal women with Cystic Fibrosis related Bone Disease (CFBD).

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is the most common fatal heritable disease in non-Hispanic whites; CF results in frequent lung infections, chronic inflammation and progressive lung failure. With advancements in medical care, patients with CF are living longer. The median survival of women with CF born and diagnosed in 2010 is projected to be 37 years. Patients with CF are now living long enough to develop comorbidities like Cystic Fibrosis related Bone Disease (CFBD), hypogonadism manifesting as pubertal delay, premature ovarian insufficiency or hypothalamic hypogonadism. These comorbidities in women without CF can be improved by estrogen supplementation.

It is well established that treating hypogonadal (low estrogen levels) women with estrogen can improve their bone health, slow the rate of bone loss and decrease bone turnover markers. Supplemental estrogen given to hypogonadal women can improve sexual and reproductive health including reduction of perimenopausal symptoms and improvement in sexual function which can improve quality of life. There is very little research investigating the effects of estrogen treatment for hypogonadal women with CF. The purpose of this study is to test the hypothesis that daily oral estrogen supplements given to hypogonadal women with CFBD will improve their bone health, sexual and reproductive health, and quality of life and modify markers of inflammation and lung function.

ELIGIBILITY:
Inclusion Criteria:

* Adult and adolescent female CF patients (age ≥ 18 years),
* presenting to the CF clinic for routine follow up of cystic fibrosis,
* hypogonadal women defined as E2 level < 25,
* dual energy X-ray absorptiometry (DEXA) scan within 2 years of enrollment with T- or Z-score < -1,
* able to tolerate oral medications.

Exclusion Criteria:

* Inability to obtain or declined informed consent from the subject and/or legally authorized representative,
* Pregnancy,
* Too ill to participate in study based on investigator's or study team's opinion,
* Current use of systemic estrogen,
* History of thromboembolic event within the previous 2 years,
* History of migraines with aura,
* Hypercoagulability including previous diagnosis of Factor V Leiden or Protein C or S deficiency,
* Current smoker,
* History of diagnosis with breast or uterine cancer,
* Current significant liver disease with cholelithiasis or cirrhosis,
* Status post lung or liver transplantation,
* Current use of systemic steroids

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in serum estradiol level in picograms per milliliter (pg/mL) from baseline to 6 months among the treatment and placebo groups | Baseline/Enrollment visit and at 6 months
  Serum estradiol measures the amount of the hormone estradiol in the blood. The level is measured using a blood test that is performed at baseline/enrollment visit and at 6 months. According to Mayo Medical Laboratories, normal levels of estradiol (E2) for menstruating women range from 15 to 350 picograms per milliliter (pg/mL). The levels of estradiol among both groups are recorded and compared from baseline to 6 months.

SECONDARY OUTCOMES:
Change in Serum carboxy-terminal collagen crosslinks (CTX-1) from baseline to 6 months among the treatment and placebo groups | Baseline/Enrollment visit and at 6 months
  Serum CTX is a telopeptide that can be used as a biomarker in the serum to measure the rate of bone turnover. The CTX test measures for the presence and concentration of a crosslink peptide sequence of type I collagen, found, among other tissues, in bone. This specific peptide sequence relates to bone turnover because it is the portion that is cleaved by osteoclasts during bone resorption, and its serum levels are therefore proportional to osteoclastic activity at the time the blood sample is drawn. Although laboratory normal ranges are said to be between 50 pg/mL and 450 pg/mL, serum levels in healthy patients not taking bisphosphonates tends to be above 300 pg/mL. This is measured at baseline and at 6 months between the 2 groups and compared.
change in of Serum Procollagen I Intact N-Terminal (P1NP) measured in mcg/L from baseline to 6 months among the treatment and placebo groups | Baseline/Enrollment visit and at 6 months
  Procollagen type I propeptides are derived from collagen type I, which is the most common collagen type found in mineralized bone. Procollagen type I N-terminal propeptide (P1NP) is considered the most sensitive marker of bone formation and it is particularly useful for monitoring bone formation therapies and antiresorptive therapies. It is measured through a blood test. Blood is drawn at baseline and at 6 months among the participants of both groups and compared. Reference Values for Adult male: 22-87 mcg/L; Adult female premenopausal: 19-83 mcg/L; Adult female postmenopausal: 16-96 mcg/L.
Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory score from baseline to 6 months among the treatment and placebo groups | Baseline/Enrollment visit and at 6 months
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a validated patient-reported outcome (PRO) containing both generic scales and scales specific to cystic fibrosis (CF). The CFQ-R measures functioning in a variety of domains, including Physical Functioning, Vitality, Health Perceptions, Respiratory Symptoms, Treatment Burden, Role Functioning, Emotional Functioning, and Social Functioning. Each CFQ-R domain yields standardized scores ranging from 0 to 100; higher domain scores indicate better health-related quality of life. The study aims to look at the changes in CFQ-R-Respiratory scores among the two groups. The questionnaire is administered at baseline and at follow up visits. The change in score from Baseline to 6 months is recorded and compared.
Change in percentage of FEV1 from baseline to 6 months among the treatment and placebo groups | Baseline/Enrollment visit and at 6 months
  FEV1 measures the lung functioning among the Cystic Fibrosis patients. Spirometry is used for measurement of FEV1.Spirometry is performed by deeply inhaling and forcefully exhaling into a spirometer (the device that records the various measurements of lung function). Forced expiratory volume-one second (FEV1) is a measure of how much air can be exhaled in one second following a deep inhalation. In normal people the Percentage of predicted FEV1 value is 80% or greater. 60%-69% are moderately abnormal; 35%-49% severely abnormal and less than 35% very severely abnormal. In cystic fibrosis patients it is usually less than normal. The test is administered at baseline and at follow up visits. The change in score from Baseline to 6 months is recorded and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Vin Tangpricha, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Wu M, Tirouvanziam R, Arora N, Tangpricha V. Findings from a feasibility study of estradiol for hypogonadal women with cystic fibrosis-related bone disease. Pilot Feasibility Stud. 2021 Aug 19;7(1):160. doi: 10.1186/s40814-021-00897-x. PMID 34412687